CLINICAL TRIAL: NCT04377061
Title: Clinical Characteristics and Pathogenic Mechanisms of Anemia in Non-celiac Wheat Sensitivity Compared to Celiac Disease and Irritable Bowel Syndrome
Brief Title: Anemia in Non-celiac Wheat Sensitivity
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Principal Investigator, University of Palermo
Other Study IDs: ACPM25
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Non-celiac Gluten Sensitivity; Anemia
Keywords: Non-celiac Gluten Sensitivity; Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NCWS retrospective and prospective patients: The clinical charts of NCWS patients, diagnosed by DBPC gluten/wheat challenge, between January 2001 and December 2019, attending the Department of Internal Medicine at the University Hospital of Palermo, the Department of Internal Medicine of the Hospital of Sciacca, and the Department of Medical and Surgical Sciences of the University of Bologna, will be reviewed retrospectively. The investigators prospectively will also survey patients with functional gastroenterological symptoms according to the Rome III criteria, and a definitive diagnosis of NCWS by DBPC gluten/wheat challenge. The patients will be recruited between January 2019 and January 2022 at the same centers, and at the Internal Medicine Division of the "Cervello-Villa Sofia" Hospital of Palermo, Palermo.
  Interventions: Diagnostic Test: Evaluation of anemia
- CD retrospective and prospective control patients: To compare the presence and characteristics of anemia in NCWS patients, the clinical charts of a control group of CD patients had been randomly chosen by a computer-generated method from patients diagnosed in the same centers, during the same period (2001-2019), and age- and sex-matched with the NCWS patients. The investigators prospectively will also survey a control group of CD patients randomly chosen by a computer-generated method from subjects diagnosed in the same centers, during the same period (2019-2022), and age- and sex-matched with the NCWS patients.
  Interventions: Diagnostic Test: Evaluation of anemia
- IBS retrospective and prospective control patients: To compare the presence and characteristics of anemia in NCWS patients, the clinical charts of another control group of IBS patients had been randomly chosen by a computer-generated method from patients diagnosed in the same centers, during the same period (2001-2019), and age- and sex-matched with the NCWS patients. The investigators prospectively will also survey a control group of IBS patients randomly chosen by a computer-generated method from subjects diagnosed in the same centers, during the same period (2019-2022), and age- and sex-matched with the NCWS patients.
  Interventions: Diagnostic Test: Evaluation of anemia

INTERVENTIONS:
Diagnostic Test: Evaluation of anemia — Evaluation of anemia in NCWS patients, and in CD and IBS controls, with both retrospective and prospective method.

SUMMARY:
In recent years, a new gluten- or wheat-related disease has emerged, a condition labelled "non-celiac gluten sensitivity" (NCGS) or "non-celiac wheat sensitivity" (NCWS). This is very often a self-reported condition, since patients refer to intestinal [mainly irritable bowel syndrome (IBS)-like] and/or extra-intestinal symptoms (i.e. fatigue, headache, anemia) caused by gluten or wheat ingestion, even though they do not suffer from celiac disease (CD) or wheat allergy (WA).

Among the extra-intestinal symptoms, several studies have shown, in patients with NCWS, the presence of anemia, generally mild, often with iron or folate deficiency characteristics, but no research has ever been planned with the specific intention of analyze this particular aspect of the disease.

Therefore, the aim of the present multicentric research was to analyze, both retrospectively and prospectively, the laboratory data of NCWS patients, compared to CD and IBS controls, to identify: a) the presence, severity and morphologic characteristic of anemia; 2) possible pathogenic mechanisms.

DETAILED DESCRIPTION:
In recent years, a new gluten- or wheat-related disease has emerged, a condition labelled "non-celiac gluten sensitivity" (NCGS) or "non-celiac wheat sensitivity" (NCWS). This is very often a self-reported condition, since patients refer to intestinal [mainly irritable bowel syndrome (IBS)-like] and/or extra-intestinal symptoms (i.e. fatigue, headache, anemia) caused by gluten or wheat ingestion, even though they do not suffer from celiac disease (CD) or wheat allergy (WA).

There are conflicting data about the real mechanisms which induce symptoms in NCGS/NCWS patients after wheat ingestion. Some authors suggested a prevalent role for Fermentable Oligosaccharides-Disaccharides-Monosaccharides and Polyols (FODMAPs), rather than gluten in determining the symptoms. Other studies underlined the activation of mechanisms of both innate and acquired immunity in NCWS patients after wheat ingestion.

Given the lack of a diagnostic biomarker, NCGS/NCWS mostly remains a diagnosis of exclusion, especially respect to CD and WA, so a confirmatory test is required. The "Salerno criteria" suggested the double-blind, placebo-controlled (DBPC), cross-over, gluten/wheat challenge as the gold standard test to discriminate true NCGS/NCWS patients.

By definition, NCGS/NCWS symptoms generally occur after the ingestion of gluten/wheat, disappear within a few days of a gluten-free diet (GFD) and quickly reappear when gluten/wheat is, voluntarily or accidentally, reintroduced. However, GDF is very difficult and onerous from a social (presence of gluten in many industrial food products and "contamination", both domestic and extra-domestic), psychological (e.g. for adolescents, exclusion from the "peer group", with difficulty in accepting the diagnosis) and economic point of view.

Among the extra-intestinal symptoms, several studies have shown, in patients with NCWS, the presence of anemia, generally mild, often with iron or folate deficiency characteristics, but no research has ever been planned with the specific intention of analyze this particular aspect of the disease.

Therefore, the aim of the present multicentric research was to analyze, both retrospectively and prospectively, the laboratory data of NCWS patients, compared to CD and IBS controls, to identify: a) the presence, severity and morphologic characteristic of anemia; 2) possible pathogenic mechanisms, with particular attention to iron, vitamin B12 and folate metabolism, thyroid hormones, and autoimmune gastric involvement.

ELIGIBILITY:
Inclusion Criteria:

1. To diagnose NCWS the recently proposed criteria will be adopted. All the patients will meet the following criteria:

   - negative serum anti-transglutaminase (anti-tTG) and anti-endomysium (EmA) immunoglobulin (Ig)A and IgG antibodies, absence of intestinal villous atrophy, negative IgE-mediated immune-allergy tests to wheat (skin prick tests and/or serum specific IgE detection), resolution of the IBS symptoms on standard elimination diet, excluding wheat, cow's milk, egg, tomato, chocolate, and other self-reported food(s) causing symptoms, symptom reappearance on double-blind placebo-controlled (DBPC) wheat challenge. As the investigators previously described in other studies, DBPC cow's milk protein challenge and other "open" food challenges will be performed too.
2. To diagnose CD the standard criteria will be adopted. All the patients will meet the following criteria:

   - positive serum anti-transglutaminase (anti-tTG) and anti-endomysium (EmA) immunoglobulin (Ig)A and IgG antibodies presence of intestinal villous atrophy.
3. To diagnose IBS the standard Rome II (for retrospective patients) and Rome III (for prospective patients) Criteria will be adopted. None of these subjects improved on an elimination diet without wheat, cow's milk, egg, tomato, or chocolate.

Exclusion Criteria:

For NCWS diagnosis it will be evaluated the following exclusion criteria:

- positive EmA in the culture medium of the duodenal biopsies, also in the case of normal villi/crypts ratio in the duodenal mucosa, self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study, other previously diagnosed gastrointestinal disorders, other previously diagnosed gynaecological disorders, nervous system disease and/or major psychiatric disorder, physical impairment limiting physical activity.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will enroll NCWS patients, both with retrospective and prospective methods. As controls groups, we will enroll CD and IBS patients, both with retrospective and prospective methods.
Sampling Method: Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Presence, severity and morphologic characteristic of anemia | At baseline and at 24 months
  red blood cells (adults references ranges, RR, 4.5-5.9 million cells/mcL, men, 4.1-5.1 million cells/mcL, women), hemoglobin (RR 13-17 g/dL, men, 12-15 g/dL, women), hematocrit (RR 40%-52%, men, 36%-47%, women), mean corpuscular volume (RR 80-100 fL), mean corpuscular hemoglobin (RR 0.4-0.5 fmol/cell), mean corpuscular hemoglobin concentration (RR 30-35 g/dL), red cell distribution width (RR 11.5%-14.5%)

SECONDARY OUTCOMES:
Possible pathogenic mechanisms | At baseline and at 24 months
  reticulocytes count (RR 0.5%-1.5%), total serum iron (RR 65-180 µg/dL, men, 30-170 µg/dL, women), ferritin (RR 12-300 ng/mL, men, 12-150 ng/mL, women), transferrin (200-350 mg/dL), total iron-binding capacity (RR 45-85 µmol/L), vitamin B12 (RR 130-700 ng/L), folic acid (RR 7-36 nmol/L), thyroid-stimulating hormone (TSH, RR 2-10 μU/mL), anti-nuclear antibodies (ANA), anti-intrinsic factor (IFA) and/or parietal cell (APCA) antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Mansueto, MD, Principal Investigator — University of Palermo
Locations (3):
- Italy (3):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Internal Medicine Division of the "Cervello-Villa Sofia" Hospital, Palermo, PA
  - Department of Internal Medicine, University Hospital of Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mansueto P, Soresi M, La Blasca F, Fayer F, D'Alcamo A, Carroccio A. Body Mass Index and Associated Clinical Variables in Patients with Non-Celiac Wheat Sensitivity. Nutrients. 2019 May 29;11(6):1220. doi: 10.3390/nu11061220. PMID 31146428
- [Result] Carroccio A, Giannone G, Mansueto P, Soresi M, La Blasca F, Fayer F, Iacobucci R, Porcasi R, Catalano T, Geraci G, Arini A, D'Alcamo A, Villanacci V, Florena AM. Duodenal and Rectal Mucosa Inflammation in Patients With Non-celiac Wheat Sensitivity. Clin Gastroenterol Hepatol. 2019 Mar;17(4):682-690.e3. doi: 10.1016/j.cgh.2018.08.043. Epub 2018 Aug 21. PMID 30138736
- [Result] Carroccio A, D'Alcamo A, Cavataio F, Soresi M, Seidita A, Sciume C, Geraci G, Iacono G, Mansueto P. High Proportions of People With Nonceliac Wheat Sensitivity Have Autoimmune Disease or Antinuclear Antibodies. Gastroenterology. 2015 Sep;149(3):596-603.e1. doi: 10.1053/j.gastro.2015.05.040. Epub 2015 May 27. PMID 26026392
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Volta U, De Giorgio R, Caio G, Uhde M, Manfredini R, Alaedini A. Nonceliac Wheat Sensitivity: An Immune-Mediated Condition with Systemic Manifestations. Gastroenterol Clin North Am. 2019 Mar;48(1):165-182. doi: 10.1016/j.gtc.2018.09.012. Epub 2018 Dec 13. PMID 30711208
- [Result] Uhde M, Ajamian M, Caio G, De Giorgio R, Indart A, Green PH, Verna EC, Volta U, Alaedini A. Intestinal cell damage and systemic immune activation in individuals reporting sensitivity to wheat in the absence of coeliac disease. Gut. 2016 Dec;65(12):1930-1937. doi: 10.1136/gutjnl-2016-311964. Epub 2016 Jul 25. PMID 27459152
- [Result] Volta U, Pinto-Sanchez MI, Boschetti E, Caio G, De Giorgio R, Verdu EF. Dietary Triggers in Irritable Bowel Syndrome: Is There a Role for Gluten? J Neurogastroenterol Motil. 2016 Oct 30;22(4):547-557. doi: 10.5056/jnm16069. PMID 27426486
- [Result] Volta U, Caio G, De Giorgio R. Is Autoimmunity More Predominant in Nonceliac Wheat Sensitivity Than Celiac Disease? Gastroenterology. 2016 Jan;150(1):282. doi: 10.1053/j.gastro.2015.08.058. Epub 2015 Nov 23. No abstract available. PMID 26616572
- [Result] De Giorgio R, Volta U, Gibson PR. Sensitivity to wheat, gluten and FODMAPs in IBS: facts or fiction? Gut. 2016 Jan;65(1):169-78. doi: 10.1136/gutjnl-2015-309757. Epub 2015 Jun 15. PMID 26078292
- [Result] Di Sabatino A, Volta U, Salvatore C, Biancheri P, Caio G, De Giorgio R, Di Stefano M, Corazza GR. Small Amounts of Gluten in Subjects With Suspected Nonceliac Gluten Sensitivity: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over Trial. Clin Gastroenterol Hepatol. 2015 Sep;13(9):1604-12.e3. doi: 10.1016/j.cgh.2015.01.029. Epub 2015 Feb 19. PMID 25701700
- [Result] Caio G, Volta U, Tovoli F, De Giorgio R. Effect of gluten free diet on immune response to gliadin in patients with non-celiac gluten sensitivity. BMC Gastroenterol. 2014 Feb 13;14:26. doi: 10.1186/1471-230X-14-26. PMID 24524388